CLINICAL TRIAL: NCT03842397
Title: OPtimisation of Surgical Repair for Treating Insufficiency of the MItral Valve - Safety Evaluation (OPTIMISE)
Brief Title: OPtimisation of Surgical Repair for Treating Insufficiency of the MItral Valve - Safety Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kephalios (Industry)
Responsible Party: Sponsor
Organization: Affluent Medical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMISE
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Mitral Valve Regurgitation
Keywords: Mitral regurgitation; Mitral valve repair; Mitral annuloplasty; Adjustable annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implanted Patients (Experimental): Implantation of Kephalios Device 1
  Interventions: Device: Kephalios Device 1

INTERVENTIONS:
Device: Kephalios Device 1 — The Kephalios Device 1 is an adjustable annuloplasty ring, to be implanted by open surgery, having a hollow structure that comprises a flat rigid ring surrounding a deformable cage. The unique feature of the Kephalios Device 1 is that its annular shape and dimension can be finely adjusted percutaneously by an external actuator (three-balloon catheter) independently in the three areas corresponding to P1, P2 and P3

SUMMARY:
The optimal surgical approach in functional mitral regurgitation (MI) was questioned in favour for prosthetic replacement due to the reduced risk of recurrent MI . However, adjustable mitral rings may provide an alternative . In this first-in-man trial, a novel balloon-adjustable mitral-ring was assessed regarding clinical safety and feasibility. 5 patients will be enrolled according to the inclusion/ exclusion criteria and subsequently implanted with the study device. Study visits will be performed preoperatively, perioperatively, at discharge, at 30 days, 3 months and 6 months. Primary outcome parameter will be morbidity and mortality at 30 days following implantation.

ELIGIBILITY:
Inclusion Criteria:

Patients

1. with symptomatic severe Mitral Regurgitation (Carpentier's classification Type I or II P2) or in asymptomatic subjects with preserved Left Ventricle function and new onset of atrial fibrillation or pulmonary hypertension;
2. with EuroScore II < 4;
3. with Left Ventricle Ejection Fraction ≥ 55%;
4. with normal coronary angiogram (no significant lesions);
5. in satisfactory condition, based on the physical exam and investigator's experience, with a life expectancy above one year after the intervention;
6. willing to sign the informed consent;
7. willing to undergo all medical follow-up, echocardiography examinations and laboratory tests planned for the clinical investigation.

Exclusion Criteria:

Patients

1. of age < 18 years;
2. who are pregnant;
3. nursing mothers;
4. who require undergoing MRI examination;
5. involved in any other clinical investigation for drugs or devices;
6. with previous cardiac surgery or diaphragmatic lesion or previous hepatic surgery;
7. needing acute intervention;
8. with active endocarditis (or having had active endocarditis in the last three months);
9. with active myocarditis;
10. with heavily calcified mitral annulus or mitral valve anatomy with a high risk of valve replacement instead of valve repair;
11. needing any cardiac surgery other than mitral repair, tricuspid valve annuloplasty, pacemaker implantation (epicardial), exclusion of left appendage (with device or surgically) and Maze (or PVI) procedure;
12. with severe pulmonary hypertension (systolic pulmonary artery pressure at rest >65 mmHg);
13. with LV Ejection Fraction < 55%;
14. with creatinine level > 2.0 mg/100ml;
15. with echocardiographic measurements predicting SAM (see specific echocardiography protocol);
16. unable to take anticoagulation medications;
17. with a known untreatable allergy to contrast media or nickel;
18. with a major or progressive non-cardiac disease that, in the investigator's experience, results in a life expectancy shorter than 1 year, or for whom the implant of the device produces an unacceptable increase of risk;
19. having had an acute preoperative neurological deficit, myocardial infarction, or cardiac event that has not returned to baseline or stabilized ≥ 30 days prior to the planned surgical procedure.
20. unable to understand and sign the ICF in absence of legal protection
21. unable to read and write
22. anticipated ring size very small (26mm) or very large (36mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety of the Kephalios Device 1 in terms of mortality | 30 days after implant
  Valve-relatedness determined according to the STS/AATS/EACTS report - Akins, C. W., Miller, D. C., Turina, M. I., Kouchoukos, N. T., Blackstone, E. H., Grunkemeier, G. L., … Lytle, B. W. (2008). Guidelines for Reporting Mortality and Morbidity After Cardiac Valve Interventions. The Annals of Thoracic Surgery, 85(4), 1490-1495. https://doi.org/10.1016/j.athoracsur.2007.12.082alve-relatedness determined according to the STS/AATS/EACTS report - Akins, C. W., Miller, D. C., Turina, M. I., Kouchoukos, N. T., Blackstone, E. H., Grunkemeier, G. L., … Lytle, B. W. (2008). Guidelines for Reporting Mortality and Morbidity After Cardiac Valve Interventions. The Annals of Thoracic Surgery, 85(4), 1490-1495. https://doi.org/10.1016/j.athoracsur.2007.12.082
Assessment of the safety of the Kephalios Device 1 in terms of morbidity | 30 days after implant
  Morbid events determined according to the STS/AATS/EACTS report - Akins, C. W., Miller, D. C., Turina, M. I., Kouchoukos, N. T., Blackstone, E. H., Grunkemeier, G. L., … Lytle, B. W. (2008). Guidelines for Reporting Mortality and Morbidity After Cardiac Valve Interventions. The Annals of Thoracic Surgery, 85(4), 1490-1495. https://doi.org/10.1016/j.athoracsur.2007.12.082

SECONDARY OUTCOMES:
Safety in terms of mortality | 3 and 6 months after implant
  Valve-relatedness determined according to the STS/AATS/EACTS report - Akins, C. W., Miller, D. C., Turina, M. I., Kouchoukos, N. T., Blackstone, E. H., Grunkemeier, G. L., … Lytle, B. W. (2008). Guidelines for Reporting Mortality and Morbidity After Cardiac Valve Interventions. The Annals of Thoracic Surgery, 85(4), 1490-1495. https://doi.org/10.1016/j.athoracsur.2007.12.082
Safety in terms of morbidity | 3 and 6 months after implant
  Morbid events determined according to the STS/AATS/EACTS report - Akins, C. W., Miller, D. C., Turina, M. I., Kouchoukos, N. T., Blackstone, E. H., Grunkemeier, G. L., … Lytle, B. W. (2008). Guidelines for Reporting Mortality and Morbidity After Cardiac Valve Interventions. The Annals of Thoracic Surgery, 85(4), 1490-1495. https://doi.org/10.1016/j.athoracsur.2007.12.082
Effectiveness in terms of increase of mitral leaflets coaptation | in the immediate post-operative phase
  through data objectively measured through echocardiography
Effectiveness in terms of reduction of Mitral Regurgitation | in the immediate post-operative phase
  through data objectively measured through echocardiography
Effectiveness in terms of absence of recurrent Mitral Regurgitation | At hospital discharge or 30 days if subject is still hospitalized, and 6 months
  through data objectively measured through echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Martin ANDREAS, MBA,PhD, Principal Investigator — Medical University of Vienna - Department of Surgery, Division of Cardiac Surgery
Locations (1):
- Medical University of Vienna - Department of Surgery, Division of Cardiac Surgery, Vienna, Austria